CLINICAL TRIAL: NCT01195805
Title: The Effect of Amiloride and Spironolactone on Renovascular and Cardiovascular Variables in Patients With Essential Hypertension in a Doubleblinded, Randomized, Placebo-controlled, Crossover Study.
Brief Title: The Effects of Amiloride and Spironolactone on Renophysiological and Cardiovascular Variables
Acronym: hass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Erling Bjerregaard Pedersen, professor, Regional Hospital Holstebro
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: MED.RES.HOS.2010.03.SKM
Record Dates: First submitted 2010-09-03; First posted 2010-09-06 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2013-03

CONDITIONS: Essential Hypertension
Keywords: Blood pressure, PWV, HRV, PWV, potassium
MeSH Terms: conditions — Essential Hypertension | interventions — Spironolactone; Amiloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Amiloride (Active Comparator)
  Interventions: Drug: Amiloride
- Spironolactone (Active Comparator)
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): 1 tablet twice a day for 28 days
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Spironolactone — 1 tablet twice a day for 28 days
  Arms: Spironolactone
Other: Placebo — 1 tablet twice a day for 28 days
  Arms: Placebo
Drug: Amiloride — 1 tablet twice a day for 28 days
  Arms: Amiloride

SUMMARY:
The investigators wish to study the effect of retaining potassium. The participants have essential hypertension. The test substances are Amiloride, Spironolactone and placebo. The participants will ingest tablets for 28 days before being examined. We will perform a 24 hours urine collection, 24-hours bloodpressure measurement, blood and urine samples and we also examine the patient using a SphygmoCor.

DETAILED DESCRIPTION:
Purpose of the study is to examine the effect of amiloride and spironolactone on

1. Renal function (GFR, u-AQP2, u-ENaCβ, u-cAMP, u-PGE2, CH20, FENa, FEK),
2. Pulsewave velocity, augmentation index central bloodpressure,
3. Vasoactive hormones (PRC, AngII, Aldo, AVP, ANP, BNP and Endot), and
4. Ambulatory bloodpressure

ELIGIBILITY:
Inclusion Criteria:

* hypertension,
* BMI 18,5-30,
* non-smoker

Exclusion Criteria:

* Smoking
* Not using contraceptives
* Other illnesses
* Drug or alcohol abuse

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Bloodpressure | 24-hours and examination

CONTACTS AND LOCATIONS:
Overall Officials: Solveig K Matthesen, MD, Principal Investigator — Departments of medical research and medicine
Locations (1):
- Departments of medical research and medicine, Holstebro, Denmark